CLINICAL TRIAL: NCT01867229
Title: Etude Prospective Multicentrique de l'aménorrhée Chimio-induite et de sa réversibilité Dans le Cancer du Sein Chez Des Patientes préménopausées Recevant Une chimiothérapie Adjuvante ou néoadjuvante. Etude Améno-Chimio.
Brief Title: Breast Cancer and Chemo-amennorhea
Acronym: chemo-ameno
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: UCL-gyneco-001; 2009/07DEC/377 (Other: CEHF)
Record Dates: First submitted 2013-05-29; First posted 2013-06-03 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer
Keywords: pre-menauposal; neo-adjuvant or adjuvant chemotherapy; no metastases
MeSH Terms: conditions — Breast Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- FEC- TC: Fluorouracil- Epiadriamycine- Cyclophosphamide Taxotère-Cyclophosphamide
  Interventions: Other: observational

INTERVENTIONS:
Other: observational — standard of care fore patients with non metastatic breast cancer

SUMMARY:
Relation between chemotherapy and amennorhea

ELIGIBILITY:
Inclusion Criteria:

pre-menauposal breast cancer needed to be treat with chemotherapy -

Exclusion Criteria:

metastases menopausal

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: pre-menauposal breast cancer treated with chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2011-10; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
incidence and duration of the amenorrhea induced by chemotherapy | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: jean-Pascal Machiels, Principal Investigator — UCL-Saint Luc
Locations (6):
- Belgium (5):
  - Clinique Saint Vincent, Rocourt, Liège
  - Cliniques Universitaires Saint-Luc, Brussels
  - Centre Hospitalier Université de Liège, Liège
  - CHR Citadelle, Liège
  - Centre hospitalier Peltzer La Tourelle, Verviers
- Institut Claudius Renaud, Toulouse, France